CLINICAL TRIAL: NCT06270563
Title: High Intensity Laser Therapy Versus Scapular Stabilization Exercises on Ventilatory Function in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Mohamed Elsadany, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003967
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Forward Head Posture
Keywords: High Intensity Laser Therapy; Scapular Stabilization Exercises; Ventilatory Function; Forward Head Posture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): They received postural advice and traditional exercise treatment (stretching and strengthening exercises) for 3 times per week for 12 weeks.
  Interventions: Other: Postural advice; Other: Traditional exercise treatment
- Group B (Experimental): They received postural advice, traditional exercise treatment (stretching and strengthening exercises), and scapular stabilization exercises 3 times per week for 12 weeks.
  Interventions: Other: Postural advice; Other: Traditional exercise treatment; Other: Scapular stabilization exercises
- Group C (Experimental): They received postural advice, traditional exercise treatment (stretching and strengthening exercises), and high intensity laser therapy 3 times per week for 12 weeks.
  Interventions: Other: Postural advice; Other: Traditional exercise treatment; Other: High intensity Laser therapy

INTERVENTIONS:
Other: Postural advice — The patients received advice about maintaining good posture when sitting, standing, reading, driving, or lifting; taking breaks; sleeping on back or side with a pillow supporting head/neck; avoiding prolonged phone use; adjusting car seat; reading stand for upright posture; keeping objects close when lifting; and using pillows for support when breastfeeding.
Other: Traditional exercise treatment — The exercise program included strengthening of deep flexor muscles and shoulder retractors while stretching of cervical extensors and pectoral muscles.
Other: Scapular stabilization exercises — Scapular Stabilization exercise was composed of four exercise programs, including scapula retraction exercise, scapula mobilization exercise, and scapula dynamic stabilization exercise I and II.
  Arms: Group B
Other: High intensity Laser therapy — There were two phases in every session, the wavelength is 1064 nm, size of spacer is 60 mm in both phases:
  Phase I (analgesic phase): the application was made by moving the applicator perpendicular to the skin in continuous circular movements at trigger points detected by acupuncture, power was 8.00 w with a dosage of 5 J/cm2, surface area 50 cm2, frequency 25 HZ, treatment time in this phase was 3 minutes and total energy received at this phase was 250 J.
  Phase II (bio stimulation): the application was made at the pain inflicting region by using continuous linear movements and prevent static application, The power was 8.00 w with a continuous frequency, dosage of 50 J/cm2, surface area 50 cm2, treatment time in this phase was 5 minutes and the total energy that was delivered to the patient during this phase was 2500 J.
  Arms: Group C

SUMMARY:
The purpose of the study is to compare between the efficacy of high intensity LASER therapy and scapular stabilization exercises on ventilatory functions in forward head posture patients

DETAILED DESCRIPTION:
Neck pain is a common complaint in the population, with a considerable impact on individuals and their families, communities, health-care systems and businesses. The estimated 1-year incidence of neck pain ranges between 10.4 and 21.3%, and the overall prevalence of neck pain in general population can be as high as 86.8%.

The photothermic and the photochemical effects of high intensity LASER therapy may increase blood flow and stimulate collagen production within tendons; in addition, high intensity LASER therapy may increase vascular permeability and has an anti-inflammatory effect, thus removing the pain stimulus.

Scapular stabilization exercise is used as an effective way to recover the imbalance in posture and the muscles. It is also effective in increasing muscle activation in the serratus anterior and lower trapezius, through decreasing the compensatory movement, which is caused by the forward head posture, and in decreasing muscle activation on the upper trapezius. Furthermore, it brings about a spinal curve change and upper crossed syndrome improvement.

Therefore, this study will compare the difference between the effect of high intensity laser therapy and scapular stabilization as a modality of treatment on ventilatory function in forward head posture patients.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages ranged from 30 -40 years.
2. All patients were diagnosed with forward head posture. - Diagnostic criteria for forward head posture by craniovertebral angle that detected by radiography and was less than 49° using specific goniometer.
3. Patients with abnormal values of decreased Forced vital capacity (FVC), forced expiratory volume at one second (FEV1), FEV1/FVC, MVV and TLC due to forward head posture.
4. All patients are medically and psychologically stable
5. They had a score more than 40% at neck disability index.

Exclusion Criteria:

1. Patients who had congenital anomalies in the neck and the thoracic cage.
2. Patients with pulmonary diseases (with restrictive lung disease or with obstructive lung disease).
3. Patients with BMI > 30 kg/m2.
4. patients with Contraindications for HILT: malignancies and potential precancerous growths, patients with cochlear implants, endocrine glands disease, patients with febrile conditions, epilepsy, pregnancy, freckles or tattoos, photosensitive medication.
5. Uncontrolled diabetes.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 12 weeks
  It was assessed by a spirometer before and after treatment. The patient was asked to breath 3 tidal breaths then fully expire, then take a deep inspiration to expire forcefully and rapidly as much as possible through the mouthpiece, the procedure was repeated 3 times and the best record was taken.
Forced expiratory volume at one second (FEV1) | 12 weeks
  It was assessed by a spirometer before and after treatment. The patient was asked to breath 3 tidal breaths then fully expire, then take a deep inspiration to expire forcefully and rapidly as much as possible through the mouthpiece, the procedure was repeated 3 times and the best record was taken.
FEV1/FVC | 12 weeks
  The ratio between the forced expiratory volume at one second (FEV1) and forced vital capacity (FVC) was calculated before and after treatment.
Maximum voluntary ventilation (MVV) | 12 weeks
  It was assessed by a spirometer before and after treatment. The patients were instructed to breathe rapidly and deeply for 15 to 30 seconds, ventilatory volumes were recorded, and the maximal volume achieved over 15 consecutive seconds was expressed in liters per minute.
Craniovertebral angle (CVA) | 12 weeks
  It was measured by a specific goniometer that was positioned parallel to the C7 Spinous process and the goniometer's movable arm on the anterior cartilage of the ear. The angle between the movable arm and the perpendicular line passing through the C7 vertebrae was recorded.
Neck Disability Index (NDI) | 12 weeks
  It is a ten-item questionnaire that was used to assess disability associated with neck pain and whiplash. There are four items that relate to subjective symptomatology (pain intensity, headache, concentration, sleeping) and six items that relate to activities of daily living (lifting, work, driving, recreation, personal care, reading).

SECONDARY OUTCOMES:
Upper thoracic chest expansion | 12 weeks
  It was measured using a tape measure at the axillary level before and after treatment.
Middle thoracic chest expansion | 12 weeks
  It was measured using a tape measure at the nipple level before and after treatment.
Lower thoracic chest expansion | 12 weeks
  It was measured using a tape measure at the level of the tip of the xiphoid process before and after treatment.
Visual analogue scale (VAS) | 12 weeks
  It was used to assess neck pain intensity; it is graded scale from 10 to 0 at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Akram A. Sayed, Prof., Study Chair — Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Cairo University, Giza, Egypt